CLINICAL TRIAL: NCT00536770
Title: A Randomized Phase 2 Study of Gemcitabine ± Erlotinib and DN-101 Versus Gemcitabine ± Erlotinib and Placebo in Subjects With Advanced Pancreatic Adenocarcinoma
Brief Title: A Study of Gemcitabine ± Erlotinib and DN-101 Versus Gemcitabine ± Erlotinib and Placebo in Patients With Advanced Pancreatic Cancer
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: DSMB
Sponsor: Novacea (Industry)
Collaborators: Schering-Plough (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 011-017
Record Dates: First submitted 2007-09-26; First posted 2007-09-28 (Estimated); Last update posted 2007-11-06 (Estimated); Status verified 2007-11

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Erlotinib Hydrochloride; Calcitriol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- A (Placebo Comparator): Placebo + gemcitabine
  Interventions: Drug: Placebo + gemcitabine
- B (Placebo Comparator): Placebo + gemcitabine + erlotinib
  Interventions: Drug: placebo + gemcitabine + erlotinib
- C (Active Comparator): DN-101 + gemcitabine
  Interventions: Drug: calcitriol + gemcitabine
- D (Active Comparator): DN-101 + gemcitabine + erlotinib
  Interventions: Drug: calcitriol + gemcitabine + erlotinib

INTERVENTIONS:
Drug: placebo + gemcitabine + erlotinib
  Arms: B
Drug: Placebo + gemcitabine
  Arms: A
Drug: calcitriol + gemcitabine
  Arms: C
Drug: calcitriol + gemcitabine + erlotinib
  Arms: D

SUMMARY:
The purpose of this study is to determine the safety and efficacy of an investigational study drug DN-101 (calcitriol) when given in combination with gemcitabine ± erlotinib in the treatment of pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of locally advanced and unresectable, or metastatic pancreatic cancer
* Performance status 0, 1,or 2
* Adequate bone marrow, renal and hepatic function

Exclusion Criteria:

* Prior chemotherapy or radiation therapy for pancreatic cancer
* Prior treatment for other cancers in last 6 months
* Cancer of the brain or spine
* Active uncontrolled infection
* Hypercalcemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2007-09

PRIMARY OUTCOMES:
Overall survival rate at 6 months

SECONDARY OUTCOMES:
Objective response rate
Duration of progression free survival
Duration of overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Novacea Investigational Site, Nashville, Tennessee, United States